CLINICAL TRIAL: NCT02772484
Title: An Evaluation of Non-invasive ICP Monitoring in Patients Undergoing Routine Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HeadSense Medical (Industry)
Collaborators: State Medical Center, Republic of Armenia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-032
Record Dates: First submitted 2016-05-12; First posted 2016-05-13 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Stroke
Keywords: noninvasive monitoring
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HS-1000 recording (Experimental): The recording session should be performed in a quiet environment with no disturbance to the patient for a total of up to 60 minutes.
  Interventions: Device: HS-1000

INTERVENTIONS:
Device: HS-1000

SUMMARY:
The HS-1000 device, an investigational intracranial monitoring device, has the potential to safely and quickly diagnose and assess stroke (and potentially other neurologic conditions) with minimal discomfort to patients. HS-1000 has the capability to establish cerebral hemodynamic measurements in suspected stroke within minutes, assist with appropriate management of stroke, and also provide an objective diagnostic tool for clinicians to monitor recovery.

DETAILED DESCRIPTION:
A prospective study will be conducted on patients with suspected stroke and/or acute neurologic changes treated at the Armenia Republican Medical Center. Male and Female patients over the age of 18 will be eligible for enrollment into the study. Eligible patients or their legally authorized representative (LAR) will be approached for consent to participate in the study. An initial recording session using the HeadSense HS-1000 device will be obtained upon admission to the hospital. During the admission, 2-4 additional recording sessions with the HS-1000 will be completed.

The end-point of the study is to collect up to 30-minute recording with up to 5 sessions of adequate quality for analysis from up to 200 subjects. This data will be correlated with clinical findings obtained during the patient's diagnosis and treatment course. An ease-of-use questionnaire will be administered to the HS-1000 device operator(s) to obtain information regarding the function and workflow aspects of using the HS-1000 in an acute setting to improve assessment, diagnosis and treatment after stroke. The data obtained from the HS-1000 recordings will be analyzed to establish specific waveform patterns correlated with brain physiology after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, > 18 years of age
* Subjects with suspected stroke and/or acute neurologic changes admitted to Armenia Republican Medical Center
* Subject or legally authorized representative (per local regulation) is able and willing to comply with the requirements of the protocol
* Subject or legally authorized representative (per local regulation) is able to understand and sign written informed consent to participate in the study

Exclusion Criteria:

* Local ear infection
* Known allergy or hypersensitivity to any of the test materials or contraindication to test materials
* Subjects currently enrolled in or less than 30 days post-participation in other investigational device or drug study(s), or receiving other investigational agent(s)
* Any condition that may jeopardize study participation (e.g., abnormal clinical or laboratory finding) or interpretation of study results, or may impede the ability to obtain informed consent (e.g., mental condition)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of HS recordings that correlate with clinical findings in the diagnosis of stroke | 60 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Ara Ghazaryan, Principal Investigator — State Medical Center, Republic of Armenia
Locations (1):
- State Medical Center, Republic of Armenia, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No